CLINICAL TRIAL: NCT06919276
Title: Longitudinal Patterns of Non-Combustible Tobacco Product Use in Adolescents (EPIC) / Assessing Development Patterns of Vaping, Alcohol, Nicotine, and Cannabis Use and Emotional Well-being (ADVANCE)
Brief Title: Nicotine and Cannabis Vape Labeling Experiment - Spring 2025
Acronym: EPIC/ADVANCE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Adam Leventhal, University Professor of Population & Public Health Sciences and Psychology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UP-23-00483/HS-19-00682; 5K24DA048160 (NIH); 5U54CA180905-12 (NIH); 5R01CA229617-06 (NIH)
Record Dates: First submitted 2025-02-28; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Vaping; Adolescent; Electronic Cigarette Use; Nicotine; Cannabis
Keywords: vaping device; product labeling; use susceptibility; perceived harm; nicotine; cannabis
MeSH Terms: conditions — Vaping; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of seven labeling conditions and one of three device colors/flavors.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (21):
- Mint - Labeling Condition 1 (Experimental): Participants will view an image of a mint-colored and flavored vape with label condition 1.
  Interventions: Other: Vaping Device Labeling
- Mint - Labeling Condition 2 (Experimental): Participants will view an image of a mint-colored and flavored vape with label condition 2.
  Interventions: Other: Vaping Device Labeling
- Mint - Labeling Condition 3 (Experimental): Participants will view an image of a mint-colored and flavored vape with label condition 3.
  Interventions: Other: Vaping Device Labeling
- Mint - Labeling Condition 4 (Experimental): Participants will view an image of a mint-colored and flavored vape with label condition 4.
  Interventions: Other: Vaping Device Labeling
- Mint - Labeling Condition 5 (Experimental): Participants will view an image of a mint-colored and flavored vape with label condition 5.
  Interventions: Other: Vaping Device Labeling
- Mint - Labeling Condition 6 (Experimental): Participants will view an image of a mint-colored and flavored vape with label condition 6.
  Interventions: Other: Vaping Device Labeling
- Mint - Labeling Condition 7 (Experimental): Participants will view an image of a mint-colored and flavored vape with label condition 7.
  Interventions: Other: Vaping Device Labeling
- Original - Labeling Condition 1 (Experimental): Participants will view an image of a white colored and original vape with label condition 1.
  Interventions: Other: Vaping Device Labeling
- Original - Labeling Condition 2 (Experimental): Participants will view an image of a white colored and original vape with label condition 2.
  Interventions: Other: Vaping Device Labeling
- Original - Labeling Condition 3 (Experimental): Participants will view an image of a white colored and original vape with label condition 3.
  Interventions: Other: Vaping Device Labeling
- Original - Labeling Condition 4 (Experimental): Participants will view an image of a white colored and original vape with label condition 4.
  Interventions: Other: Vaping Device Labeling
- Original - Labeling Condition 5 (Experimental): Participants will view an image of a white colored and original vape with label condition 5.
  Interventions: Other: Vaping Device Labeling
- Original - Labeling Condition 6 (Experimental): Participants will view an image of a white colored and original vape with label condition 6.
  Interventions: Other: Vaping Device Labeling
- Original - Labeling Condition 7 (Experimental): Participants will view an image of a white colored and original vape with label condition 7.
  Interventions: Other: Vaping Device Labeling
- Blueberry - Labeling Condition 1 (Experimental): Participants will view an image of a blue-colored and blueberry flavored vape with label condition 1.
  Interventions: Other: Vaping Device Labeling
- Blueberry - Labeling Condition 2 (Experimental): Participants will view an image of a blue-colored and blueberry flavored vape with label condition 2.
  Interventions: Other: Vaping Device Labeling
- Blueberry - Labeling Condition 3 (Experimental): Participants will view an image of a blue-colored and blueberry flavored vape with label condition 3.
  Interventions: Other: Vaping Device Labeling
- Blueberry - Labeling Condition 4 (Experimental): Participants will view an image of a blue-colored and blueberry flavored vape with label condition 4.
  Interventions: Other: Vaping Device Labeling
- Blueberry - Labeling Condition 5 (Experimental): Participants will view an image of a blue-colored and blueberry flavored vape with label condition 5.
  Interventions: Other: Vaping Device Labeling
- Blueberry - Labeling Condition 6 (Experimental): Participants will view an image of a blue-colored and blueberry flavored vape with label condition 6.
  Interventions: Other: Vaping Device Labeling
- Blueberry - Labeling Condition 7 (Experimental): Participants will view an image of a blue-colored and blueberry flavored vape with label condition 1.
  Interventions: Other: Vaping Device Labeling

INTERVENTIONS:
Other: Vaping Device Labeling — Participants will view one vape image (experimental stimulus) and are randomized to a label presented and the color/flavor of the vaping device presented.
  The label conditions are:
  1. plain (i.e., no labeling on device)
  2. "contains THC"
  3. "contains 80% THC"
  4. "contains 80% THC - HIGH POTENCY"
  5. "contains nicotine"
  6. "contains 5% nicotine"
  7. "contains 5% nicotine - HIGH STRENGTH" The color/flavor conditions are: mint/mint, white/original, blue/blueberry.

SUMMARY:
This study assesses how the ways in which nicotine and cannabis vaping devices are labeled impact use susceptibility, anticipated effects, and health harm.

DETAILED DESCRIPTION:
The primary objectives of the study: (1) Determine whether different device labels with the contained substance (nicotine or cannabis) affect adolescent use susceptibility, anticipated effects or impairment, and perceived health harms; (2) Determine whether device color/product flavor differentially impact the study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be enrolled in a partnering high school.

Exclusion Criteria:

* Participants who cannot independently understand study consent and the study surveys are ineligible.

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3900 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Use Intention Susceptibility | 5 minutes
  This 3-item self-report measure assesses participant interest in trying the vaping device in the future. A 4-level Likert scale is used: definitely not, probably not, probably yes, definitely yes.
Perceived Health Harms | 5 minutes
  This 2-item self-report measure assesses participant perception of health harms and risks associated with using the vaping product. A 4-level Likert scale is used: definitely not, probably not, probably yes, definitely yes.
Anticipated Subjective Effects | 5 minutes
  This 9-item self-report measure assesses anticipated subjective effects from using the vaping device. Participants will select all that apply.
Anticipated Impairment/Enhancement | 5 minutes
  This 4-item self-report measure assesses participant anticipated enhancement or impairment effects on completing different activities due to using the vaping product. A 5-level Likert scale is used: definitely make it harder, probably make it harder, no effect, probably make it easier, definitely make it easier.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No